CLINICAL TRIAL: NCT02194400
Title: A Double-Blind, Placebo-Controlled Dose Escalation Study of the Administration of Multiple Intravenous Doses of RSLV-132 in Subjects With Systemic Lupus Erythematosus
Brief Title: Dose Escalation Study of RSLV-132 in Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Resolve Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132-02
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: RSLV-132; Systemic Lupus Erythematosus; Lupus; SLE; Resolve
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — RSLV-132

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Saline infusion
  Interventions: Biological: RSLV-132
- RSLV-132 (Experimental): 0.3 - 10 mg/kg experimental drug
  Interventions: Biological: RSLV-132

INTERVENTIONS:
Biological: RSLV-132 — 0.3 - 10.0 mg/kg RSLV-132 weekly for 4 weeks

SUMMARY:
A one month multi-dose study will evaluate the safety and tolerability of 3 intravenous infusions of RSLV-132 in subjects with inactive to mild SLE.

ELIGIBILITY:
Inclusion Criteria:

* Stable SLE with no anticipated change in medications for the next 60 days

Exclusion Criteria:

* Other biologic drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James Posada, Ph.D., Study Chair — Resolve Therapeutics
Locations (4):
- United States (4):
  - Clinical Research of West Florida, Clearwater, Florida
  - West Michigan Rheumatology, Grand Rapids, Michigan
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research, Dallas, Texas

REFERENCES:
- See also: Resolve Therapeutics Website — http://www.resolvebio.com
- See also: Lupus Research Institute — http://www.lupustrials.org